CLINICAL TRIAL: NCT04344015
Title: Collection of COVID-19 Convalescent Plasma
Brief Title: COVID-19 Plasma Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20D.346
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma Donation (Other): The goal of this study is to identify individuals who have previously been infected with COVID-19 and collect plasma from those who meet inclusion criteria for convalescent plasma donation. This protocol will allow for the collection, manufacturing, and storage of convalescent plasma that may be administered to patients with COVID-19 in the near future. In addition, it allows for testing of SARS-COV-2 antibody titers in the plasma that has been collected to inform studies assessing outcomes for patients currently infected with COVID-19 who have received convalescent plasma infusions.
  Interventions: Other: Plasma Donation

INTERVENTIONS:
Other: Plasma Donation — Previously infected COVID-19 patients will be recruited to donate convalescent plasma.

SUMMARY:
Patients who are severely ill with COVID-19 may benefit from receiving plasma infusions from donors who have recovered from the disease and are proven to no longer be infected. Efforts to initiate the collection and infusion of these products to high risk patients have been initiated around the world and the FDA has recently provided information about how this could be accomplished. As the Jefferson Blood Donor Center already has processes to collect, test and process blood, investigators are planning to make efforts to collect plasma for this use should it be necessary. The purpose of this study is to describe the process for identifying and collecting convalescent plasma from donors previously infected with the virus. The research portion on top of this standard blood product collection will the process of identification of subjects and processes by which blood products are processed in this special population. This protocol does not involve the administration of blood products to patients with COVID-19 infection.

DETAILED DESCRIPTION:
As described by the FDA on 3/24/2020, convalescent plasma has been used for a variety of infectious diseases including Ebola, SARS, MERS and H1N1 flu. Given that there is no current medical treatment beyond supportive care for COVID-19, there is a great deal of interest in using convalescent plasma for patients with COVID-19. As a first step in this process, investigators are proposing to identify donors and collect plasma with antibodies against COVID-19. While the intention is to use this for patients in the near future, the purpose of this study will be to see if this is feasible and a separate application will be submitted related to the treatment of patients with these products.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Prior diagnosis of COVID-19 documented by a laboratory test approved by the FDA
* Either: Complete resolution of all COVID-related symptoms for 14-28 days at the time of blood donation AND negative repeated SARS-CoV-2 test OR Complete resolution of all COVID-related symptoms for > 28 days
* Male donors, never-pregnant female donors, or previously pregnant female donors negative for HLA antibodies
* Meet all criteria for volunteer blood donation per Jefferson Blood Donor Center and the FDA

Exclusion Criteria:

* Failure to pass standard volunteer blood donor screening criteria required by the Jefferson Blood Donor Center and the FDA
* Female donors with HLA antibodies (per FDA requirements for convalescent plasma donors)
* Inadequate venous access for phlebotomy
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Number of patients who screen eligible for donation | 1 year
  # of individuals screened eligible
Number of patients who consent to plasma donation | 1 year
  # of patients who consent to donation
Number of plasma donations received | 1 year
  # of plasma donations received

SECONDARY OUTCOMES:
Safety of donation procedures | 1 year
  Side effects or adverse events related to plasma donation

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States